CLINICAL TRIAL: NCT07020910
Title: The Bad Berka Heart Rhythm Registry (2B2R) is a Prospective, Single-center Observational Cohort Evaluating Safety, Efficacy, and Outcomes in Patients Undergoing Arrhythmia Therapy or CIED Implantation at the Heart Center Bad Berka
Brief Title: Bad Berka Heart Rhythm Registry of Patients With or at Risk of Arrhythmias Treated at Heart Center Bad Berka
Acronym: 2B2R
Status: Recruiting | Type: Observational
Sponsor: Zentralklinik Bad Berka (Other)
Responsible Party: Principal Investigator, Santi Raffa, Dr. PhD., Zentralklinik Bad Berka
Other Study IDs: # 23333/2024/62
Record Dates: First submitted 2025-05-22; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Arrhythmias
Keywords: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Bad Berka Heart Rhythm Registry (2B2R) is a prospective, single-center observational cohort designed to systematically collect and analyze data of patients undergoing cardiac arrhythmia therapy as well as implantation of cardiac electronic devices (CIEDs) at the Heart Center Bad Berka.

The register aims to evaluate procedural safety, acute and long-term efficacy, and clinical outcomes across a broad spectrum of arrhythmias and interventional strategies, including novel technologies such as pulsed field ablation (PFA) and conduction system pacing. The registry is intended to generate real-world evidence to support clinical decision-making, identify predictors of outcomes, and contribute to quality assurance and innovation in the field of cardiac electrophysiology.

DETAILED DESCRIPTION:
The field of cardiac electrophysiology continues to evolve rapidly, with new tools and techniques improving both arrhythmia diagnosis and therapy. While randomized controlled trials provide critical insights, real-world data from clinical practice are essential to evaluate safety, efficacy, and long-term outcomes across diverse patient populations and treatment modalities.

The 2B2R registry aims to bridge this gap by collecting comprehensive clinical data of patients referred for cardiac arrhythmia treatment including drug therapy, electrophysiological studies, catheter ablation (e.g. atrial fibrillation, atrial flutter, atrial and AV-node dependent supraventricular tachycardia, premature ventricular contractions, and ventricular tachycardia), interventional stroke-prevention, as well as device implantation at the Heart Center Bad Berka.

Data will be prospectively collected, procedural parameters, complication rates, acute success, follow-up outcomes, imaging, device therapy, and patient-reported outcomes will be assessed. Substudies focused on specific arrhythmias or technologies (e.g., pulsed field ablation, high-density mapping, or device therapy such as conduction system pacing) will be embedded within the registry.

The data will be analyzed to: - Evaluate clinical effectiveness and safety of interventional EP procedures - Assess predictors of arrhythmia recurrence or procedural complications - Compare technologies and procedural strategies

- Monitor quality metrics and inform continuous process improvement Participation in the registry does not influence clinical management which remains at the discretion of the treating physicians. The registry complies with all applicable data protection and ethical standards.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* At risk of or with documented cardiac arrhythmia undergoing medical or interventional therapy at the Heart Center Bad Berka
* Informed consent obtained

Exclusion Criteria:

* Inability or unwillingness to provide informed consent
* Participation in another interventional trial that precludes registry inclusion

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Cardiac Arrhythmias or at Risk for the Development of Cardiac Arrhythmias Undergoing Drug-Therapy or Interventional Procedures at the Heart Center Bad Berka
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2034-08-01 (Estimated)

PRIMARY OUTCOMES:
Acute Treatment Success | Perioperative/Periprocedural
  1. Acute Treatment Success Defined as acute symptom control and achievement of predefined procedural endpoints (e.g. AV-nodal modification, elimination of accessory pathway conduction, pulmonary vein isolation, bidirectional block across linear ablation lesions, suppression of ectopic beats, non-inducibility of the clinical arrhythmia, effective occlusion of the left atrial appendage, successful CIED-implantation)
Safety (peri-procedural Complications) | within 30 days
  Incidence of major complications (e.g. development of ventricular proarrhythmia, tamponade, stroke, vascular injury, AV-block, phrenic nerve palsy, pneumothorax, hemothorax, lead dislodgment, or death)

SECONDARY OUTCOMES:
Arrhythmia Recurrence | through study completion, an average of 1 year
  Documented recurrence of the treated arrhythmia after the blanking period (if applicable), using scheduled 24-48h Holter-ECG, 12-lead-ECG, CIEDs, and smart devices (e.g. smart-watch…).
All-cause Rehospitalization | through study completion, an average of 1 year
  Number of hospitalizations following the index procedure.
Symptom and Quality of Life Improvement | through study completion, an average of 1 year
  Based on structured follow-up or telephone follow up where applicable.
Device Therapy Outcomes (in patients with CIEDs)- 1.Lead performance - | through study completion, an average of 1 year
  evaluation of implanted cardiac device leads (pacemaker, ICD, CRT) in terms of electrical integrity, sensing and pacing thresholds, impedance stability.
Device Therapy Outcomes (in patients with CIEDs) - 2. Appropriate and inappropriate therapies- | through study completion, an average of 1 year
  Number and type of appropriate and inappropriate device therapies (e.g., anti-tachycardia pacing or shocks) delivered by implantable cardioverter-defibrillators (ICDs) or CRT-Ds.
Device Therapy Outcomes (in patients with CIEDs)-3. Device related complications- | through study completion, an average of 1 year
  Incidence of device-related complications following implantation of cardiac implantable electronic devices (CIEDs), including lead dislodgement, infection, hematoma requiring intervention, pneumothorax, lead fracture, insulation failure, and pocket erosion.

CONTACTS AND LOCATIONS:
Locations (1):
- Zentralklinik Bad Berka, Bad Berka, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Keelani A, Alothman O, Borisov G, Frommhold M, Bartoli L, Abdelwahab H, D'Ambrosio G, Shehri SA, Raffa S, Geller JC. Feasibility and Clinical Efficacy of Focal Pulsed Field Ablation in Patients With Non-Pulmonary Vein Triggered Atrial Arrhythmia From the Superior Caval Vein. J Cardiovasc Electrophysiol. 2025 Feb;36(2):359-366. doi: 10.1111/jce.16510. Epub 2024 Dec 10. PMID 39654529